CLINICAL TRIAL: NCT00007917
Title: A Phase I Trial Of Gemcitabine Followed By Flavopiridol In Patients With Solid Tumors
Brief Title: Gemcitabine Plus Flavopiridol in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-166; U01CA062490 (NIH); P30CA006516 (NIH); DFCI-00166; NCI-24; CDR0000068344 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-01-06; First posted 2003-10-15 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — alvocidib; Gemcitabine

ARMS (1):
- Arm I (Experimental): Patients receive gemcitabine IV over 1-2.5 hours on days 1 and 8 and flavopiridol IV continuously over 24 hours on days 2 and 9. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of gemcitabine and flavopiridol until the maximum tolerated dose (MTD) is reached. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Drug: alvocidib; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: alvocidib
Drug: gemcitabine hydrochloride

SUMMARY:
Phase I trial to study the effectiveness of gemcitabine plus flavopiridol in treating patients who have advanced solid tumors. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of gemcitabine and flavopiridol in patients with advanced solid tumors.

II. Determine the toxicity and safety profile of this regimen in these patients.

III. Determine the pharmacokinetic profile of this regimen in this patient population.

OUTLINE: This is a dose-escalation study.

Patients receive gemcitabine IV over 1-2.5 hours on days 1 and 8 and flavopiridol IV continuously over 24 hours on days 2 and 9. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of gemcitabine and flavopiridol until the maximum tolerated dose (MTD) is reached. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 6-58 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven solid tumor for which gemcitabine is a treatment option or for which no effective therapy exists
* Previously untreated disease allowed
* No large and potentially symptomatic pericardial effusion or undrained pleural effusion (with or without pleurodesis)
* No CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 2,000/mm3
* Platelet count at least 100,000/mm3
* No prior thrombotic events

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 2 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No clinically significant cardiac disease
* No prior deep venous thrombus
* No prior arterial vascular event
* No prior myocardial infarction
* No unstable angina
* No prior transient ischemic attack or cerebrovascular accident
* No cardiac arrhythmias that could be related to cardiac ischemia

Pulmonary:

* No clinically significant pulmonary disease
* No history of pulmonary embolism

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection
* No severe malnutrition or intractable emesis
* No chronic diarrheal disease within the past 6 months

PRIOR CONCURRENT THERAPY:

Chemotherapy:

* No more than 1 prior chemotherapy regimen
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* Prior gemcitabine or flavopiridol allowed
* No other concurrent chemotherapy

Radiotherapy:

* At least 3 weeks since prior radiotherapy and recovered
* No prior radiotherapy to more than 50% of bone marrow
* No concurrent radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2001-01; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Shapiro, MD, PhD, Study Chair — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts